CLINICAL TRIAL: NCT01094522
Title: A Randomized, Double-blind, Controlled, Multi-site Study of the Pharmacokinetics and Pharmacodynamics of Methadone vs. Morphine During Mechanical Ventilation Following Cardiac Surgery in Neonates, Infants and Children
Brief Title: Measuring the Amount of Methadone or Morphine in the Blood of Neonates, Infants & Children After Cardiac Surgery.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Colorado, Denver (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Gregory Hammer, Professor of Anesthesia and Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-03012010-5083; IRB Protocol # 16739
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Methadone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Methadone (Experimental): One half the Study patients will be randomized to receive a loading dose of IV methadone, followed by IV doses (given by the ICU nurse), on a PRN basis, for pain control for up to 24 hours during their postoperative course while they are intubated.
  Interventions: Drug: Methadone
- Morphine (Active Comparator): One half the Study patients will be randomized to receive a loading dose of IV morphine, followed by IV doses (given by the ICU nurse), on a PRN basis, for pain control for up to 24 hours during their postoperative course while they are intubated.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — 0.2 mg/kg (IV) for the Initial Loading Dose; followed by PRN ("as needed") doses (given by the ICU Nurses) starting at 0.035 mg/kg (IV) every 30 minutes, for postoperative pain. The PRN dose of methadone may be increased by the ICU doctors until the dose is adequate to relieve the patient's pain.
  Arms: Methadone
Drug: Morphine — 0.2 mg/kg (IV) for the Initial Loading Dose; followed by PRN ("as needed") doses (given by the ICU Nurses) starting at 0.035 mg/kg (IV) every 30 minutes, for postoperative pain. The PRN dose of morphine may be increased by the ICU doctors until the dose is adequate to relieve the patient's pain.
  Other Names: MS
  Arms: Morphine

SUMMARY:
Study Population:

Neonates, infants and children from birth to 5 years of age undergoing cardiac surgery with CPB.

The use of methadone to provide analgesia may be increasing due to advantages compared to other commonly used opioid analgesic drugs. While efficacy of methadone has been reported in adults, there is a paucity of information in neonates and infants. In the latter population, fentanyl and morphine are most commonly used for opioid analgesia following major surgery, while methadone is frequently used for weaning of opioid dependent and tolerant patients, in spite of the paucity of knowledge of methadone pharmacology in this population. There are several clinical problems associated with fentanyl and morphine, and methadone may offer superior efficacy with fewer side effects than these agents. We propose to study the pharmacokinetics (PK) and pharmacodynamics (PD) of methadone in neonates and infants in the intensive care unit following cardiac surgery.

DETAILED DESCRIPTION:
Treatment:

Fentanyl will be administered for intraoperative analgesia by the treating anesthesiologist in a dose range of 25 - 50 mcg/kg. No other intraoperative opioids will be given.

Subjects will receive intravenous methadone or morphine ("study drug") delivered by an initial IV "bolus" injection followed by a nurse-administered patient controlled analgesia (PCA) device for postoperative pain for a period of 24 hours. The initial dose of study drug will be 0.2 mg/kg IV administered following admission to the ICU after surgery. The study drug will then be given at a dose of 0.035 mg/kg IV as needed q30min via PCA. The study drug may be increased or decreased in increments of 20-25% according to the discretion of the investigator as needed to maintain a FLACC pain assessment tool < 4. Subjects will also receive lorazepam 0.025 mg/kg IV q2hr as needed for agitation as indicated by specific criteria. The study drug will be discontinued after 24 hours to facilitate "wash out" sampling and determination of elimination half-life. Beginning at 24 hours, fentanyl will be used for analgesia at an equianalgesic dose to be determined by the investigator based upon the current PCA "study drug" dose.

Measurements and Monitoring:

* Blood samples will be obtained for measurement of concentrations of methadone (methadone group) and morphine and its metabolites, morphine-3-glucuronide and morphine-6-glucuronide (morphine group), prior to administration of initial bolus dose (t = 0) and t = 5 min, 15 min, 30 min, 60 min, 2 hrs, 4 hrs and 6 hrs; thereafter, blood samples will be obtained for measurement every 6 hrs for up to 90 hrs according to availability of vascular access for phlebotomy.
* Continuous monitoring: temperature (rectal), electrocardiogram, heart rate, systemic arterial blood pressure, central venous blood pressure, respiratory rate, oxygen saturation (pulse oximetry)
* Intermittent recording (q1hr): urine output
* Lab Tests (at baseline[prior to study procedures] and 24 hours after initial dose of study medication): arterial blood gas tensions, arterial lactate, Hb/Hct, BUN/Cr, glucose, AST, ALT
* 12 lead ECG at hour 24 for determination of QTc.
* The Faces, Legs, Activity, Cry, Consolability (FLACC) Scale recoded every hour, and preceding every study medication PCA dose for 24 hours.
* Subject follow up at 90 hours to record time of extubation, re-intubation if necessary, and reason for re-intubation.

Primary Endpoints: Pharmacokinetics of methadone and morphine, including its metabolites (morphine-3-glucuronide and morphine-6-glucuronide)

Secondary Endpoints:

* Pain scores (FLACC) during the 24 hours study period
* Amount of study drug administered during the 24-hour dosing period
* Changes in heart rate, systemic arterial blood pressure and laboratory test values

ELIGIBILITY:
Inclusion Criteria:

Neonates, infants and children from birth through 5 years of age undergoing mechanical ventilation following cardiac surgery for congenital heart disease. Congenital heart lesions include "two ventricle repairs", including tetralogy of Fallot, transposition of the great arteries, "unobstructed" total anomalous pulmonary venous return, truncus arteriosus, atrioventricular canal defect and ventricular septal defect.

Exclusion Criteria:

Subjects will be excluded from the study because of prematurity (gestational age < 37 weeks), weight < 3.0 kg, severe hepatic dysfunction (elevation of conjugated bilirubin > 2, AST/ALT > 200 IU/L), significant renal dysfunction (serum Cr > 1.5 mg/dL), participation within 30 days of study entry or within 5 times the half-life, whichever is longer, in another investigational drug study, or previous participation in this study. Patients will be excluded if they have received opioids for more than 12 hours of the 48-hour period prior to surgery. In addition, patients will be excluded if they have a history of other clinically significant medical problems, which, in the opinion of the investigator, would interfere with study participation.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hammer, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado, Denver, Colorado
  - Oregon Health & Sciences University, Portland, Oregon

REFERENCES:
- [Result] Ward RM, Drover DR, Hammer GB, Stemland CJ, Kern S, Tristani-Firouzi M, Lugo RA, Satterfield K, Anderson BJ. The pharmacokinetics of methadone and its metabolites in neonates, infants, and children. Paediatr Anaesth. 2014 Jun;24(6):591-601. doi: 10.1111/pan.12385. Epub 2014 Mar 26. PMID 24666686
- [Result] Elkomy MH, Drover DR, Glotzbach KL, Galinkin JL, Frymoyer A, Su F, Hammer GB. Pharmacokinetics of Morphine and Its Metabolites in Infants and Young Children After Congenital Heart Surgery. AAPS J. 2016 Jan;18(1):124-33. doi: 10.1208/s12248-015-9826-5. Epub 2015 Sep 9. PMID 26349564

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 47 subjects were enrolled. 7 were withdrawn prior to randomization. 40 were randomized.
Period: Overall Study
Arm/Group | Methadone | Morphine
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone | Morphine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 1.00 [0.01 to 3.79] | 1.37 [0.01 to 5.39] | 1.19 [0.01 to 5.39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration of Morphine Including Its Metabolites (Morphine-3-glucuronide and Morphine-6-glucuronide)
Time Frame: 0, 15, 30 minutes, 1, 2, 4, 6 hrs, every 6 hrs up to 24 hrs
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Morphine
Number analyzed (Participants) | 20
ng/mL
  Morphine | 27.55 [0.317 to 348]
  M3G | 225 [0.39 to 2630]
  M6G | 22.95 [0.861 to 383]

2. Secondary Outcome: •Pain Scores (FLACC) During the 24 Hours Study Period
Description: Average of hourly FLACC score for each subject over 24 hours was calculated, followed by median and full range for total subjects in each arm.
  FLACC (Face, Leg, Activity, Cry, Consolability) score ranges from 0-10 with 0 representing no pain
Time Frame: 24 hours
Population: Hourly FLACC score was calculated for 16 subjects in Methadone group and 19 subjects in morphine group
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Methadone | Morphine
Number analyzed (Participants) | 16 | 19
units on a scale | 1.375 [0 to 3.375] | 1.917 [0 to 4.792]

3. Secondary Outcome: •Amount of Study Drug Administered During the 24-hour Dosing Period
Time Frame: 24 hours
Measure: Mean (Full Range); unit: mg
Arm/Group | Methadone | Morphine
Number analyzed (Participants) | 20 | 20
mg | 8.56 [1 to 29.4] | 13.77 [1.7 to 88.7]

4. Primary Outcome: Maximum Concentration of Methadone Including Its Metabolites (EDDP and EMDP)
Time Frame: 0, 15, 30 minutes, 1, 2, 4, 6 hrs, every 6 hrs up to 24 hrs
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Methadone
Number analyzed (Participants) | 20
ng/mL
  Methadone | 52.35 [0.702 to 829]
  EDDP | 3.42 [0.257 to 108]
  EMDP | 0.194 [0.101 to 0.537]

ADVERSE EVENTS:
Arm/Group | Methadone | Morphine
Serious Adverse Events (participants affected / at risk) | 5/20 | 3/20
Other Adverse Events (participants affected / at risk) | 5/20 | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone (N=20) | Morphine (N=20)
Culture negative sepsis (Infections and infestations) | 1 (1) | 0 (0)
Left vocal cord paralysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Left pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema requiring re-intubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure requiring re-intubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 1 (1) | 0 (0)
Duodenal atresia requiring surgery (Gastrointestinal disorders) | 0 (0) | 1 (1)
Apnea requiring re-intubation (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone (N=20) | Morphine (N=20)
Self-extubation (Investigations) | 0 (0) | 2 (2)
Culture negative sepsis (Infections and infestations) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema requiring re-intubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 1 (1) | 0 (0)
Duodenal atresia requiring surgery (Gastrointestinal disorders) | 0 (0) | 1 (1)
Apnea requiring re-intubation (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No